CLINICAL TRIAL: NCT02950844
Title: Identification, Electro-mechanical Characterisation and Ablation of Driver Regions in Persistent Atrial Fibrillation (STAR MAPPING)
Brief Title: Identification, Electro-mechanical Characterisation and Ablation of Driver Regions in Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011040; PG/16/10/32016 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Electrogram; Ablation; Drivers
MeSH Terms: conditions — Atrial Fibrillation

ARMS (1):
- STAR mapping guided ablation (Experimental): Patients will undergo PVI guided ablation in addition to STAR mapping guided ablation. The impact on electrophysiological endpoints including cycle length prolongation and AF termination will be assessed.
  Interventions: Other: Novel mapping algorithm

INTERVENTIONS:
Other: Novel mapping algorithm — Mapping and ablation of atrial fibrillation drivers identified by the STAR mapping algorithm.
  In a sub-study a novel mapping system (CARTOFINDER, Biosense Webster, Inc, CA) was used in mapping drivers in AF.
  Other Names: STAR MAPPING

SUMMARY:
Atrial fibrillation (AF) is the most common sustained heart rhythm abnormality. Its incidence is increasing partly due to the ageing population and it has been referred to as a growing epidemic. AF results in irregular contractions of the heart causing unpleasant symptoms of palpitations and increasing the risk of stroke, heart failure and death. Percutaneous catheter ablation is a safe treatment option in symptomatic patients with AF. The success rate of these procedures have improved with time due to our better understanding of AF, development of new techniques and technology, and greater physician experience. However, the success rate of these procedures still only remains around 70%. This is contributed to our limited ability to find the areas that drive the AF.

STAR mapping is a novel mapping system that has been developed with a view of better identifying the sites that drive AF, through taking into account the mechanisms of AF that have already been demonstrated. Data from this study will be used to refine the identification of drivers in the fibrillation left atrium with enormous potential to simplify ablation and improve success rates and thereby reducing the need for further procedures.

To better validate this mapping system the investigators also aim to use it in participants with atrial tachycardia (AT), which is a heart rhythm abnormality of which the mechanism can be readily identified with the existing mapping systems used in clinical practice. The investigators will demonstrate that the STAR mapping algorithm can effectively map AT.

To gain further understanding of the changes that occur in the left upper chamber of the heart in the context of AF half of the participants with AF will undergo cardiac magnetic resonance imaging to assess for the presence of scar. This will enhance our understanding of how atrial remodelling promotes AF, which may point to ways of modifying this process and preventing AF.

DETAILED DESCRIPTION:
AF catheter ablation success rates are still limited to around 70% with a large proportion of patients requiring to have further procedures to remain in normal heart rhythm. The current strategies that are used in catheter ablation of AF involve targeting the pulmonary veins that enter the left sided upper chamber of the heart. The supportive evidence in targeting other areas beyond the pulmonary veins remains mixed. Thereby with the existing mapping systems other sites that potentially drive AF have not been effectively identified. Further to this, it has also been suggested that these sites are intermittent and mobile in nature making it more difficult to effectively map. With this in mind the investigators have developed STAR mapping, a novel mapping system that takes these factors into account. The purpose of this study is to use this mapping system prospectively to effectively map and ablate drivers of AF as identified by termination and/or slowing of AF during the catheter ablation.

Participants that have documented AF that has been present all the time for less than 24 months i.e. early persistent AF and that have been referred for catheter ablation for AF by an Electrophysiologist will be recruited into the study.

Participants will undergo consenting for the procedure and their involvement in the research study. The procedures will be conducted either under local anaesthetic/sedation or general anaesthetic depending on the clinical needs of the patient. During the procedure tubes will be passed into the left upper chamber of the heart through the groin. Through these tubes catheters will be used to create a geometry of the heart chamber. Following this, in half of the participants a basket catheter with 64 electrodes will be positioned in the upper chamber whilst conventional catheters will be used in the other half of the participants. This is to demonstrate that this mapping system can effectively be used with a variety of mapping catheters. The signals collected will then be used in the novel mapping system to identify sites as potential drivers of AF. These sites will then be targeted and the response to ablation will be recorded particularly looking at slowing and/or termination of the AF, which will support these sites identified as drivers.

As part of the validation phase of the study participants that have been scheduled for a catheter ablation for AT by their Electrophysiologist will be enrolled into the study. The STAR maps generated in these cases will be compared to the maps generated by the conventional system. This will enable validation of the STAR mapping system.

The mapping system used for this study will be CARTOFINDER (CARTO, Biosense Webster, Inc, CA). Analyses using this mapping system will allow a sub-study on identifying mechanisms of AT and drivers in AF using the CARTOFINDER system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to provide informed consent
2. Patients with AT (whether de novo or occuring post AF ablation) undergoing catheter ablation (validation phase)
3. Patients with early persistent AF <24months undergoing their first catheter ablation (mapping phase)

Exclusion Criteria:

1. Unwillingness to sign consent
2. Age <18 years old
3. Contraindications for catheter ablation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with AT that have STAR maps that are consistent with conventional maps. | During the catheter ablation
  The number of participants with AT that have STAR maps acquired with multi-polar mapping catheters (basket or other) that yield consistent maps with mechanisms corresponding to those identified by conventional mapping.
Number of participants with AF that have STAR maps that suggest a small number of drivers sustain AF. | During the catheter ablation
  The number of participants with consecutive STAR maps acquired with multi-polar mapping catheters (basket or other) that demonstrate a consistent proportion of wave fronts with a given activation pattern suggesting a small number of drivers (whether consistent or intermittent) sustaining AF.
Number of participants with AF and AT that have an ablation effect. | During the catheter ablation
  The number of participants that had a response to ablation (slowing or termination of AT/AF) that is consistent with the mechanism of AT/AF identified by the STAR mapping.

SECONDARY OUTCOMES:
The number of driver sites that correlate with sites of scar. | 30 min up to 1 hour (CMR) and during study
  The number of driver sites identified on the STAR map that correlate to sites of late gadolinium enhancement on the cardiac magnetic resonance imaging and areas of low voltage on the voltage map.
The number of sites in the left atrium with altered conduction that correlate with sites of scar. | During the catheter ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Heart Centre, London, United Kingdom

REFERENCES:
- [Derived] Honarbakhsh S, Schilling RJ, Finlay M, Keating E, Hunter RJ. Prospective STAR-Guided Ablation in Persistent Atrial Fibrillation Using Sequential Mapping With Multipolar Catheters. Circ Arrhythm Electrophysiol. 2020 Oct;13(10):e008824. doi: 10.1161/CIRCEP.120.008824. Epub 2020 Sep 9. PMID 32903033
- [Derived] Honarbakhsh S, Hunter RJ, Ullah W, Keating E, Finlay M, Schilling RJ. Ablation in Persistent Atrial Fibrillation Using Stochastic Trajectory Analysis of Ranked Signals (STAR) Mapping Method. JACC Clin Electrophysiol. 2019 Jul;5(7):817-829. doi: 10.1016/j.jacep.2019.04.007. Epub 2019 May 8. PMID 31320010